CLINICAL TRIAL: NCT04065633
Title: A PHASE 1, OPEN LABEL, SINGLE-DOSE, CROSSOVER STUDY TO EVALUATE THE BIOEQUIVALENCE OF A COMMERCIAL TABLET FORMULATION OF PF-04965842 RELATIVE TO THE PHASE III TABLET FORMULATION UNDER FASTING CONDITIONS AND THE EFFECT OF FOOD ON THE RELATIVE BIOAVAILABILITY OF THE COMMERCIAL TABLET FORMULATION IN HEALTHY PARTICIPANTS
Brief Title: Study of Commercial and Phase 3 of PF-04965842 Formulations, Estimation of Effect of Food on Commercial Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B7451032
Record Dates: First submitted 2019-07-16; First posted 2019-08-22 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Dermatitis, Atopic
Keywords: Phase 1 Bioequivalence Study; Healthy Participants; Estimation of the Effect of Food; Relative Bioavailability
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 randomized, open label, single-dose, crossover study in healthy participants to estimate the rBA of the commercial formulation of PF-04965842 (Test formulation 1) and the variant formulation with slower dissolution (Test formulation 2) compared to the Phase 3 formulation (Reference formulation), to demonstrate the BE of the commercial formulation relative to the Phase 3 formulation, and to estimate the effect of food on the rBA of the commercial formulation after a single 200 mg oral dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A sequence 1 (Experimental)
  Interventions: Drug: P3-Fast; Drug: Comm-Fast; Drug: Vari-Fast; Drug: Comm-Fed
- Part A sequence 2 (Experimental)
  Interventions: Drug: P3-Fast; Drug: Comm-Fast; Drug: Vari-Fast; Drug: Comm-Fed
- Part B sequence 1 (Experimental)
  Interventions: Drug: P3-Fast; Drug: Comm-Fast
- Part B sequence 2 (Experimental)
  Interventions: Drug: P3-Fast; Drug: Comm-Fast

INTERVENTIONS:
Drug: P3-Fast — 200 mg (2 × 100 mg) PF-04965842 Phase 3 tablet formulation under fasted conditions
Drug: Comm-Fast — 200 mg PF-04965842 commercial tablet formulation under fasted conditions
Drug: Vari-Fast — 200 mg PF-04965842 variant tablet formulation with slower dissolution under fasted conditions
  Arms: Part A sequence 1; Part A sequence 2
Drug: Comm-Fed — 200 mg PF-04965842 commercial tablet formulation under fed conditions
  Arms: Part A sequence 1; Part A sequence 2

SUMMARY:
Part A

* To measure and compare the amount of study drug in the blood after a single 200 mg dose of study drug given as the commercial tablet formulation and the Phase 3 tablet formulation under fasting conditions
* To measure and compare the amount of study drug in the blood after a single 200 mg dose given as the variant Phase 3 tablet formulation and the Phase 3 tablet formulation under fasting conditions
* To estimate the effect of food on the amount of study drug in the blood after a single 200 mg dose of the commercial formulation

Part B

• To measure and compare the amount of study drug in the blood after a single 200 mg dose given as the commercial tablet formulation and the Phase 3 tablet formulation under fasting conditions

Parts A & B

* To collect samples for genotyping (CYP2C19 and CYP2C9 - enzymes that metabolize [break down] certain medications)

  o Genotyping is the collection of a small sample of blood that contains your genes
* To evaluate the safety and tolerability of the study drug after single 200 mg doses of the three different formulations given to healthy participants
* To measure the amount of study drug in the blood after single doses of the different formulations
* To collect exploratory samples for biobanking o Biobanking is the collection and storage of blood samples for possible future testing

DETAILED DESCRIPTION:
The purpose of this study in healthy participants is to estimate the bioavailability (BA) of the commercial formulation of PF-04965842 and a variant formulation with slower dissolution relative to the Phase 3 formulation, to demonstrate the bioequivalence (BE) of the commercial formulation relative to the Phase 3 formulation, and to estimate the effect of food on the BA of the commercial formulation. This study consists of 2 parts: Part A is to estimate the relative BA (rBA) of single 200 mg doses of the commercial tablet formulation of PF-04965842 and a variant formulation of slower dissolution rate compared to the Phase 3 tablet formulation. The effect of food on the BA of the commercial tablet formulation will also be evaluated. Part B is to establish BE between the Phase 3 and commercial formulations. The study will follow a staged approach as the sample size for BE cannot be determined with currently available information.

Therefore, it is proposed to assess the maximum observed concentration (Cmax) and area under the curve (AUC) ratios between the Phase 3 and commercial formulations as well as the within-participant variability of Cmax and AUC values determined in Part A. Based on the results from Part A, the sample size of Part B will be determined and the decision to proceed to Part B will be made.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy).

  * History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis
  * Evidence or history of clinically significant dermatological condition (eg, atopic dermatitis or psoriasis) .History of tuberculosis (TB) (active or latent) or inadequately treated TB infection.
  * History of chronic infections, history of recurrent infections, history of latent infections, .History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.
  * history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Plasma PF-04965842 PK parameters | hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  AUCinf
Plasma PF-04965842 PK parameters | hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  Cmax

SECONDARY OUTCOMES:
number of subjects with treatment-emergent adverse event | baseline until Period 4 study day 35
number of subjects with significant change from baseline in Supine Blood pressure, pulse rate and oral temperature | baseline until Period 4 study day 3
  The actual and the change from baseline values will be summarized by treatment. These data will be listed and out of range values will be summarized
number of subjects with significant Changes from baseline for the ECG parameters QT interval, heart rate, QTc interval, PR | baseline until Period 4 study day 3
  Changes from baseline for the ECG parameters QT interval, heart rate, QTc interval, PR interval, and QRS complex will be summarized by treatment and time. The number (%) of participants with maximum postdose QTc values and maximum increases from baseline in the following categories will be tabulated by treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Sylvester Pawlak, APRN, Principal Investigator — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451032